CLINICAL TRIAL: NCT02011711
Title: Modulation of Mucosal and Systemic Immunity by Hormonal Contraceptives
Brief Title: Modulation of Immunity by Hormonal Contraceptives
Status: Completed | Type: Observational
Sponsor: Thomas L. Cherpes (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Thomas L. Cherpes, Assistant Professor, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 2013H0235; R01HD072663 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mirena: Women interested in beginning use of Mirena
- Depot-medroxyprogesterone acetate: Women interested in beginning use of depot-medroxyprogesterone acetate
- Oral Contraception: Women interested in beginning use of oral contraception

SUMMARY:
Clinical study to determine if hormonal contraceptive use effects cells that fight infection (i.e., immune cells).

DETAILED DESCRIPTION:
Feminization of the HIV pandemic is impetus for better understanding of the risk factors promoting male to female sexual transmission. One putative risk factor is hormonal contraceptive use. Our laboratory recently reported that dendritic cell activation, virus-specific T cell expansion, and memory T cell development were impaired among female mice administered depot-medroxyprogesterone acetate (DMPA) prior to viral infection of mucosal tissue, and we now are enrolling women into a clinical investigation exploring the immunomodulatory effects of several common hormonal contraceptive forms. Completion of this research will provide important comparative evaluation of the capacity of these drugs to modulate host defenses combating genital tract infection, eventually supplying healthcare providers more informed recommendations regarding appropriate hormonal contraceptive choices among women at risk for acquisition of HIV.

ELIGIBILITY:
Inclusion Criteria:

* not pregnant
* regular menstrual cycle

Exclusion Criteria:

* use of oral contraceptive or Mirena in 3 months prior to enrollment
* use of depot-medroxyprogesterone acetate in 6 months prior to enrollment
* diagnosis of sexually transmitted infection in 30 days prior to enrollment
* history of cervical malignancy

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women seeking to initiate use of an oral contraceptive, depot-medroxyprogesterone acetate, or Mirena.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in ectocervical permeability | Baseline and 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Cherpes, MD, Principal Investigator — Stanford University
Locations (1):
- Edwards Building, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vicetti Miguel RD, Hendricks RL, Aguirre AJ, Melan MA, Harvey SA, Terry-Allison T, St Leger AJ, Thomson AW, Cherpes TL. Dendritic cell activation and memory cell development are impaired among mice administered medroxyprogesterone acetate prior to mucosal herpes simplex virus type 1 infection. J Immunol. 2012 Oct 1;189(7):3449-61. doi: 10.4049/jimmunol.1103054. Epub 2012 Aug 31. PMID 22942424
- [Background] Quispe Calla NE, Vicetti Miguel RD, Mei A, Fan S, Gilmore JR, Cherpes TL. Dendritic cell function and pathogen-specific T cell immunity are inhibited in mice administered levonorgestrel prior to intranasal Chlamydia trachomatis infection. Sci Rep. 2016 Nov 28;6:37723. doi: 10.1038/srep37723. PMID 27892938
- [Result] Quispe Calla NE, Ghonime MG, Cherpes TL, Vicetti Miguel RD. Medroxyprogesterone acetate impairs human dendritic cell activation and function. Hum Reprod. 2015 May;30(5):1169-77. doi: 10.1093/humrep/dev035. Epub 2015 Mar 3. PMID 25740884
- [Result] Quispe Calla NE, Vicetti Miguel RD, Boyaka PN, Hall-Stoodley L, Kaur B, Trout W, Pavelko SD, Cherpes TL. Medroxyprogesterone acetate and levonorgestrel increase genital mucosal permeability and enhance susceptibility to genital herpes simplex virus type 2 infection. Mucosal Immunol. 2016 Nov;9(6):1571-1583. doi: 10.1038/mi.2016.22. Epub 2016 Mar 23. PMID 27007679
- [Result] Quispe Calla NE, Vicetti Miguel RD, Trout W, Cherpes TL. HIV and Hormonal Contraception: Bench and Bedside. J Acquir Immune Defic Syndr. 2017 Mar 1;74(3):e85-e86. doi: 10.1097/QAI.0000000000001174. No abstract available. PMID 27599006